CLINICAL TRIAL: NCT07085221
Title: Digital Out-of-hospital Management on Clinical Outcomes in Patients With Early Cardiogenic Shock: a Multi-center, Randomized Controlled Clinical Trial
Brief Title: Digital Out-of-hospital Management on Clinical Outcomes in Patients With Early Cardiogenic Shock
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Chen Jing, Chief of Cardiology Department, Renmin Hospital of Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: WDRY2024-K234
Record Dates: First submitted 2025-07-14; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2024-10

CONDITIONS: Shock, Cardiogenic; Shock
MeSH Terms: conditions — Shock, Cardiogenic; Shock

STUDY DESIGN:
Intervention Model Description: Experimental group: digital out-of-hospital management Control group: routine outpatient follow-up
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional management group (No Intervention)
- hospital external management (Experimental)
  Interventions: Combination Product: hospital external management

INTERVENTIONS:
Combination Product: hospital external management — (I) Symptom management: After enrollment, health managers regularly promoted health education to enhance patients' awareness of the disease and adherence to post-discharge management. Simultaneously, patients were managed via a digital platform, with each patient being provided with a chip-implanted sphygmomanometer to monitor their blood pressure and pulse in real time. If patients develop symptoms, they can report them in real-time and generate alerts to health managers. Through internal clinical decision-making algorithms, the telemedicine team would conduct clinical evaluations and seek decision guidance from clinical cardiologists if necessary.
  (II) Clinical evaluation: the system stratified patients by risk levels and determined the frequency and intensity of management accordingly, with blood pressure and heart rate monitored daily. The digital management system automatically transmitted abnormal data to a doctor's assistant, with early detection of life-threatening complication
  Arms: hospital external management

SUMMARY:
This clinical study was a multi-center, open-label, randomized controlled clinical trial. A total of 472 patients with early-stage cardiogenic shock were recruited and randomly divided into the experimental group and the control group, with 236 cases in each group. The HeartMed-HF digital out-of-hospital management was used to manage the patients in the experimental group, while the patients in the control group were managed according to the discharge guidance. The primary endpoints were 1-year all-cause mortality and unplanned readmission after randomization (excluding emergency department visits). Secondary endpoints (at 3 months, 6 months, and 12 months post-randomization) were: all-cause mortality, rehospitalization for HF, recurrent MI, ischemia-driven repeat revascularization, stroke, BARC 3-5 grade major bleeding, unplanned formal rehospitalization, types of GDMT medications or GDMT target dose achievement rate.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years old;
2. The patient meets the diagnosis of early-stage cardiogenic shock, with SCAI stage A, B, or C during hospitalization; (1) SCAI stage A:

Without signs of shock and meeting one of the following criteria:

1. Combined with extensive myocardial infarction, diagnosed as widespread anterior wall myocardial infarction based on ST-segment elevation in ECG leads (V1-V5, aVL, I leads), inferior wall combined with right ventricular (II, III, aVF, V3R-V5R leads) and/or posterior wall myocardial infarction (V7-V9 leads), or recurrent myocardial infarction within 28 days.
2. Concurrent acute heart failure or acute exacerbation of chronic heart failure. (2) SCAI stage B-C (meeting the following conditions)

1) 60 < SBP < 90 mmHg or mean arterial blood pressure 50 < MAP < 60 mmHg or a decrease of > 30 mmHg from baseline lasting 30 minutes; or SBP ≥ 90 mmHg but heart rate /SBP > 1 lasting > 30 minutes.

2) The highest arterial blood lactate during hospitalization < 5 mmol/L. 3. Stable clinical symptoms at discharge, defined as:

1. SBP ≥ 90 mmHg when vasoactive drugs are not used;
2. No signs and symptoms of shock. 4. Understand and be willing to sign the informed consent, and be willing to follow the treatment and visit plan required by the protocol.

Exclusion Criteria

1. Unable to use a smartphone for out-of-hospital management despite training
2. The reasons for discharge were treatment withdrawal and transfer to another hospital for continued therapy
3. Previous or current hospital admission due to cardiac arrest
4. Refractory cardiogenic shock
5. Refractory Heart Failure (ACC/AHA guidelines Stage D heart Failure)
6. Left ventricular ejection fraction < 30%
7. (Estimated) glomerular filtration rate < 25 ml/min or on dialysis
8. Severe hepatic insufficiency (Child-Pugh class C)
9. Severe chronic obstructive pulmonary disease (confirmed by pulmonary function tests, or requiring long-term home oxygen therapy or long-term use of corticosteroids)
10. History of cardiac surgery
11. Pregnant or lactating women
12. Combined with malignant tumors and other serious diseases, the expected life span is less than 1 year
13. Neuropsychiatric disorders, unable to cooperate with management;
14. Participation in other clinical trials within the past year;
15. Other circumstances considered to be inappropriate for this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year all-cause mortality and unplanned formal readmission after randomization (excluding emergency department visits) | From enrollment to the end of management up to 12 months

SECONDARY OUTCOMES:
all-cause mortality | From enrollment to the end of management up to 12 months
Rehospitalization for HF | From enrollment to the end of management up to 12 months
Recurrent MI | From enrollment to the end of management up to 12 months
Ischemia-driven repeat revascularization | From enrollment to the end of management up to 12 months
Stroke | From enrollment to the end of management up to 12 months
Bleeding Academic Research Consortium 3-5 grade | From enrollment to the end of management up to 12 months
  BARC Bleeding Classification
  • Type 0
  No evidence of bleeding.
  • Type 1
  Mild bleeding requiring no medical intervention (e.g., patient self-discontinues medication without seeking medical attention).
  • Type 2
  Overt bleeding necessitating medical intervention (e.g., medication adjustment, hospitalization, or evaluation) but not meeting criteria for higher grades.
  Examples: Subcutaneous bruising, epistaxis, or minor gastrointestinal bleeding.
  * Type 3
  * 3a: Hemoglobin drop of 3-5 g/dL or requiring transfusion;
  * 3b: Hemoglobin drop ≥5 g/dL, cardiac tamponade, need for surgical hemostasis, or vasoactive drugs;
  * 3c: Intracranial hemorrhage or intraocular bleeding causing visual impairment.
  * Type 4
  CABG-related bleeding (e.g., postoperative reoperation or massive transfusion).
  * Type 5
  * 5a: Clinically suspected fatal bleeding
Unplanned formal rehospitalization | From enrollment to the end of management up to 12 months
Types of GDMT medications | From enrollment to the end of management up to 12 months
GDMT target dose achievement rate | From enrollment to the end of management up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No